CLINICAL TRIAL: NCT07005258
Title: Evaluation of the Diagnostic Performance of the CandID PLUS PCR for the Detection of Candida Spp. in Peritoneal Fluid of Critically Ill Patients With Suspected Intra-abdominal Candidiasis
Brief Title: Diagnostic Performance of the CandID PLUS PCR for the Diagnosis of Intra-abdominal Candidiasis in Critically Ill Patients
Acronym: CANDIDIAG
Status: Completed | Type: Observational
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Sponsor
Other Study IDs: 2025PI060
Record Dates: First submitted 2025-06-03; First posted 2025-06-05 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-04

CONDITIONS: Intra-Abdominal Infection; Candida; Peritonitis Infectious; Molecular Diagnostic; Critically Ill Intensive Care Unit Patients
Keywords: intra-abdominal candidiasis; secondary peritonitis; candida; PCR; molecular diagnostic
MeSH Terms: conditions — Intraabdominal Infections; Torulopsis; Peritonitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Peritoneal fluid samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Critically ill patients with intra-abdominal candidiasis requiring abdominal surgery: All patients have confirmed intra-abdominal candidiasis (positive Candida culture)

SUMMARY:
Invasive candidiasis are the most common form of fungal infection in critically ill patients, particularly intra-abdominal candidiasis (IAC), which is associated with high morbidity and mortality. The current diagnostic gold standard relies on conventional fungal culture, which has a long turnaround time and may delay targeted antifungal therapy. Non-culture-based assays such as 1,3-β-D-glucan lack specificity for early and definitive diagnosis. Molecular diagnostics, including PCR, offer faster and more specific detection, but their clinical use remains limited.

The CandID PLUS PCR assay targets major Candida species and has not yet been evaluated on peritoneal fluid.

The CANDIDIAG study aims to assess the feasibility and diagnostic performance of the CandID PLUS PCR in detecting Candida spp. in peritoneal fluid from ICU patients with suspected IAC.

This study constitutes a post-hoc analysis of the pBDG2 study (Prospective evaluation of the peritoneal 1.3 Beta-D-glucan for the diagnosis of intra-abdominal candidiasis in the critically ill patients) registered with the number NCT 03997929). Therefore, all patients have been already recruited. For the CANDIDIAG study, we will use the biological collection of peritoneal fluid issue from the pBDG2 study. All patients with confirmed intra-abdominal candidiasis are identified. We will test de CandID PCR, retrospectively, on their peritoneal fluid and compared the results with the fungal culture.

ELIGIBILITY:
Inclusion Criteria:

* adult critically ill patient
* with confirmed intra-abdominal candidiasis (culture positive with Candida albicans, glabrata, parapsilosis, tropicalis, krusei, and dubliniensis)
* enrolled in the pBDG2 study (NCT 03997929)
* intra-abdominal candidiasis documented at

Exclusion Criteria:

* Declined to participate
* intra-abdominal candidiasis caused by other candida species

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The pBDG2 study enrolled 199 ICU patients across four participating centers. Inclusion criteria were: adult ICU patients with suspected intra-abdominal infection likely due to Candida spp., requiring emergency abdominal surgery.
  Among the enrolled patients, 88 were diagnosed with confirmed intra-abdominal candidiasis based on positive fungal culture.
  Only these 88 patients will be eligible for inclusion in the CANDIDIAG study. This constitutes a post-hoc analysis of a predefined subpopulation from the pBDG2 cohort.
  Participating centers included the University Hospitals of Nancy, Dijon, Strasbourg, and the Regional Hospital Center of Metz (CHR Metz)
Sampling Method: Non-Probability Sample
Enrollment: 88 (Actual)
Dates: Start 2025-04-17 (Actual); Primary Completion 2025-04-17 (Actual); Study Completion 2025-04-17 (Actual)

PRIMARY OUTCOMES:
To evaluate the diagnostic performance of the CandID PLUS PCR for the detection of Candida albicans, glabrata, parapsilosis, tropicalis, krusei, and dubliniensis in peritoneal fluid of ICU patients with intra-abdominal candidiasis | Day of the surgery
  Sensitivity, specificity, positive predictive value (PPV), and negative predictive value (NPV) of the CandID PLUS PCR, using fungal culture as the reference standard.

SECONDARY OUTCOMES:
To compare the diagnostic performance of the CandID PLUS PCR with that of peritoneal 1,3-β-D-glucan | Day of the surgery
  Sensitivity, specificity, PPV, and NPV of peritoneal 1,3-β-D-glucan compared with fungal culture; diagnostic performance comparison between CandID PLUS PCR and 1,3-β-D-glucan (including ROC curve analysis)
To explore the association between PCR cycle threshold (Ct) values (as a proxy for fungal load) and clinical parameters, including SOFA score and ICU mortality | Day 1 (surgery) to Day 28
  Association between PCR Ct values and clinical severity (SOFA score) and ICU mortality

CONTACTS AND LOCATIONS:
Locations (1):
- Université de Lorraine - CHRU de Nancy, Vandœuvre-lès-Nancy, Lorraine, France

IPD SHARING:
Plan to Share IPD: No